CLINICAL TRIAL: NCT00170352
Title: Hyperbaric and Normobaric Oxygen in Severe Brain Injury
Brief Title: Comparison Between Different Types of Oxygen Treatment Following Traumatic Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HSR2000-858; NIH-5 RO1 NS042126-03
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Traumatic Brain Injury
Keywords: hyperbaric oxygen; cerebral metabolism; hyperoxia; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Hyperoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Treatment (HBOT)
Procedure: Enhanced Oxygen Treatment (Enhanced FiO2)

SUMMARY:
The purpose of this study is to study the effects of EARLY (no more than 24 four hours from injury) administration of extra amounts of oxygen on traumatic brain injury.

DETAILED DESCRIPTION:
Brain injury continues to be a major cause of death and disability throughout the world. Our investigations of hyperbaric oxygen treatment (HBOT) indicate that it is a relatively safe treatment that has promise as a potential therapy for patients with severe traumatic brain injury (TBI). The goals of the present proposal are to further elucidate the mechanisms of action of HBOT on severe TBI and to test hypotheses that are crucial to the possible future design of a Phase III clinical trial.

Our initial prospective clinical trial to assess the effectiveness of HBOT in severe TBI documented very significant improvement in survival, particularly in certain subgroups of patients. In our second study, HBOT was found to improve cerebral aerobic metabolism in patients with severe TBI, reduce elevated intracranial pressure, and had a persistent positive effect for at least six hours following the treatment. Our work suggests that HBOT allows the brain to utilize increased amounts of oxygen more efficiently following treatment.

Recently, increasing the inspired oxygen concentration (FiO2) to 100% has been proposed as an alternative way of delivering supranormal levels of oxygen to severe TBI patients. Experimental investigation in the fluid percussion rat model using HBOT at 1.5 ATA (atmospheres absolute) for 60 minutes followed by 3 hours of 100%fraction of inspired oxygen (FiO2) have given optimum results in terms of mitochondrial functional and neurobehavioral improvement.

The clinical and experimental data together provide a strong basis for the restorative effect of the combination of hyper- and normobaric hyperoxia on severe TBI. The goal of this study is to evaluate the use of HBOT and 100% FiO2 separately and in combination.

ELIGIBILITY:
Inclusion Criteria:

* All closed head trauma victims with GCS score < 8, when no effects from paralytics, sedation, alcohol and/or street drugs are present.
* Informed consent obtained.
* Entry into the study within 24 hours after injury.
* If a patient enters the hospital with a mild or moderate brain injury and subsequently deteriorates to a GCS < 8 within 48 hours of admission, the patient is considered a candidate for entry into the study.
* CT scan score > II in accordance with the classification system of the Traumatic Coma Data Bank.

Exclusion Criteria:

* Consent could not be obtained.
* Patients who are brain dead or close to brain death (fixed, dilated pupils).
* Unstable pulmonary status requiring FiO2 of 50% or greater to maintain a PaO2 of 70 mm Hg or greater.
* History of severe pulmonary disease, such as COPD or asthma.
* Unstable fracture (spine, pelvis, femur, etc) preventing placement into the HBO chamber.
* Patients placed in barbiturate coma during initial management due to the potential effect barbiturates have on cerebral metabolism.
* Age range < 16 years or > 65 years.
* Coagulopathy.
* Pregnancy.
* Severe mental retardation or prior severe head injury.
* High velocity penetrating injury to the head,(e.g. gunshot wound).
* Multiple organ failure.
* Massive cerebral hemisphere or brainstem hematoma, stroke

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2002-11; Primary Completion 2007-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Cerebral Metabolic Rate of Oxygen (CMRO2)
Microdialysis Lactate
Brain tissue oxygen (PtO2)
Intracranial Pressure (ICP)

SECONDARY OUTCOMES:
Microdialysis-Glycerol,Glucose,Pyruvate,Lactate/Pyruvate Ratio
Cerebral Spinal Fluid (CSF) Lactate
Arterial-Venous Oxygen Difference (AVDO2)
Cerebral Blood Flow (CBF)
Cerebral Spinal Fluid Isoprostane
Bronchial-Alveolar Lavage Cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Gaylan L Rockswold, M.D., PhD, Principal Investigator — Hennepin County Medical Center, Minneapolis; Sarah B Rockswold, M.D., Study Director — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Rockswold SB, Rockswold GL, Zaun DA, Liu J. A prospective, randomized Phase II clinical trial to evaluate the effect of combined hyperbaric and normobaric hyperoxia on cerebral metabolism, intracranial pressure, oxygen toxicity, and clinical outcome in severe traumatic brain injury. J Neurosurg. 2013 Jun;118(6):1317-28. doi: 10.3171/2013.2.JNS121468. Epub 2013 Mar 19. PMID 23510092